CLINICAL TRIAL: NCT07058038
Title: Association of Nocturnal Hypoxemia and Benign Prostatic Hyperplasia in Patients With Obstructive Sleep Apnea
Brief Title: Nocturnal Hypoxemia and Benign Prostatic Hyperplasia in OSA Patients
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: BPH in OSA patients
Record Dates: First submitted 2025-06-27; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostate Hypertrophy(BPH), Obstructive Sleep Apnea( OSA)
Keywords: nocturnal hypoxemia- OSA-BPH
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Obstructive Sleep apnea (OSA) is a common sleep disorder characterized by frequent partial or complete obstructions of the upper airway during sleep leading to sleep fragmentation and sympathetic activation.
* The main pathophysiological findings in OSAS are due to both a dynamic obstruction of the upper airway and the fragmentation of sleep during the night. These issues result in abnormal cycles of hypoxia and re-oxygenation. This disturbance produces transient ischemia of the tissues, a concept known as chronic intermittent hypoxia (CIH) with clinical implication in several cardiometabolic diseases
* Polysomnography (PSG) is considered to be the gold standard for diagnosing sleep-related breathing disorders, which include obstructive sleep apnea (OSA), central sleep apnea, sleep-related hypoventilation disorders, and sleep related hypoxia disorder
* Benign prostate hyperplasia (BPH) is the most frequent benign neoplasm in aging men and one of the most common chronic conditions in the male population.
* Although the pathogenesis of BPH is not yet fully understood, recent evidence indicates the role of chronic inflammation in BPH, CIH which occurred in OSA patient induces systemic inflammatory processes; such chronic inflammatory conditions may contribute to tissue injury, activate cytokines release, increase the concentration of growth factors, and subsequently cause the development of BPH.
* To date, little research has focused on the relationship between OSA and BPH, especially the impact of nocturnal hypoxemia , sleep architecture ,hormonal disturbance on BPH . Therefore, the aim of our study is to illuminate association between sleep related hypoxemia and BPH in Patients with OSA

DETAILED DESCRIPTION:
All patients enrolled in the study underwent the following assessment:

1. Full History taking with stress on patient Complaint:

   Witnessed apneas during sleep. Awakening with choking or gasping sensation Loud habitual Snoring Dry mouth falling asleep during driving or motor vehicle Accidents Frequent nocturia Tiredness and Sleepiness in morning after sleep at night Awakening with a headache. Insomnia
2. Clinical examination:

   - General examination: Respiratory rate, O2 saturation, blood pressure, heart rate, lower limb edema, neck vein, thyroid enlargement, any facial deformities.
   * Anthropometric measurements:

     • Height (in meters): patients stand up straight, with buttocks, shoulder blades, and heels touching the back of the stadiometer.

     • Weight (in kilograms)
     * Body mass index (BMI) is a quantitative metric used to estimate body fat based on an individual's weight relative to height. It is calculated by dividing body weight in kilograms by the square of height in meters (BMI = weight (kg) / height² (m²).
     * Neck circumference (NC) was measured between the mid-cervical point posteriorly and mid-anterior neck (below the laryngeal prominence). Measurements were taken while the participant was standing upright and looking straight ahead)
     * Waist circumference: circumferential measurement obtained at the level of the superior iliac crest.
   * Palatine tonsil size examination

     • Size 0 (a): no visible tonsillar tissue.

     • Size 1(b): tonsils are confined within the tonsillar pillars.
     * Size 2(c): tonsils extended to the level of the pillars.
     * Size 3(d): tonsils extended beyond the pillars.
     * Size 4(e): tonsils reach the midline
   * Friedman tongue position • FTP I: the uvula and tonsils (or pillar) are fully visible • FTP IIa: most of the uvula is visible, but the tonsils/pillar are obscured • FTP IIb: the entire soft palate is visible up to the base of the uvula.

     • FTP III: only the proximal portion of the soft palate is visible, the distal end is not seen.

     • FTP IV: only the hard palate is visible, neither the uvula nor the soft palate is seen
   * Local chest examination: To exclude accompanied pulmonary diseases
3. Laboratory test

   • Complete blood count (CBC)

   • Arterial blood gases (ABG)

   • C-reactive protein (CRP).
   * Thyroid profile (TSH, T3, T4)
   * Lipid profile (Cholesterol, Triglyceride, LDL, HDL)
   * Urine analysis
   * PSA
   * Testosterone.
   * Serum Creatinine.
4. Pelviabdominal us BPH was diagnosed when there is an increase in the volume of the prostate with a calculated volume exceeding 30 mL using the formula (width x height x length x 0.52)
5. Scales & Questionnaires:

   All the questionnaires are written in English, but they were translated to Arabic for all patient and the cultural adaptation of the questions were considered.

   --Epworth sleepiness scale (ESS): The Epworth Sleepiness Scale (ESS) was used to assess the level of daytime sleepiness. In this questionnaire, participants rate their likelihood of falling asleep in various situations using a 4-point scale

   --Berlin Questionnaire: As part of the initial clinical assessment, the Berlin Questionnaire was administered to evaluate the risk of obstructive sleep apnea syndrome (OSAS). When possible, a family member or bed partner was consulted to confirm the accuracy of responses related to snoring behavior.

   --STOP-BANG score: The STOP-BANG questionnaire is one of the most widely accepted screening tools for obstructive sleep apnea (OSA).

   --International prostate symptom score: Lower urinary tract symptoms (LUTS) were assessed using the International Prostate Symptom Score (IPSS), a validated and widely used questionnaire designed to evaluate symptoms related to benign prostatic hyperplasia (BPH).
6. Polysomnography All participants underwent overnight polysomnography using the (SONMO screen plus, SOMNO medics, Germany) . Recordings were performed according to the standard montage recommended by the American Academy of Sleep Medicine (AASM). Sleep studies were scored and interpreted manually in accordance with the AASM Scoring Manual, Version 3 .

   Measured variables:

   ***Measurement of the following physiologic variables is required during polysomnography (PSG) in accordance with the latest scoring criteria of the American Academy of Sleep Medicine (AASM, 2023)

   • Sleep staging

   • Airflow
   * Respiratory effort
   * Snoring
   * Oxygen saturation
   * Electrocardiogram
   * Limb movements
   * Body position

ELIGIBILITY:
Inclusion criteria:

* Males >18 years old with symptoms suggesting obstructive sleep apnea. Exclusion criteria
* Chronic obstructive pulmonary diseases (COPD), interstitial lung disease (ILD), bronchial asthma (BA)
* Heart failure, cerebral stroke, and other severe cerebrovascular and cardiovascular diseases.
* Other sleep disorders, such as narcolepsy and restless leg syndrome, etc.
* Mixed and Central sleep apnea.
* Major mental or physical illness.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients who visited Mansoura University Hospitals sleep clinic for an initial evaluation and having symptoms consistent with sleep apnea
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
correlation between sleep related Hypoxemia and Benign Prostatic hyperplasia in Patients with OSA | 13 month
  sleep related hypoxemia can be assessed through parameters recorded during a diagnostic polysomnogram (PSG):
  * The oxygen desaturation index (ODI) : represents the number of times per hour of sleep that a patient's oxyhemoglobin saturation drops by more than a specified amount from baseline, typically 4%.
  * Mean SpO2 (%): The average oxygen saturation for the entire night.
  * T 90%: The percentage of total sleep time spent with oxygen saturation <90%.
  * Apnea hypopnea time % (AHT%): The percentage of total sleep time spent with apnea and hypopnea duration in patients with OSA

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura faculty of medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang JF, Shen N, Zhao JM, Chen ML, Wang BY, Chen GP. Relationship between severity of obstructive sleep apnea and benign prostatic hyperplasia. Sleep Breath. 2023 Mar;27(1):363-369. doi: 10.1007/s11325-022-02617-y. Epub 2022 Apr 23. PMID 35460050
- See also: Related Info — https://www.ncbi.nlm.nih.gov/sites/books/NBK558920